CLINICAL TRIAL: NCT04921020
Title: Department of Ophthalmology
Brief Title: Assessment of Eyelid Topology and Kinetics Based on Deep Learning Method
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-485
Record Dates: First submitted 2021-06-01; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Eyelid Diseases
MeSH Terms: conditions — Eyelid Diseases | interventions — Photography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Normal participants
  Interventions: Other: Photography
- Patients with blepharoptosis
  Interventions: Other: Photography
- Patients with blepharospasm
  Interventions: Other: Photography
- Patients with dry eye disease
  Interventions: Other: Photography
- Patients with Graves' disease
  Interventions: Other: Photography

INTERVENTIONS:
Other: Photography — Facial photographs and blinking videos are taken

SUMMARY:
This study plans to assess eyelid topology (such as margin reflex distance, eyelid contour, and corneal exposure area) and blinking (such as frequency, velocity, and duration), using deep learning method to automatically extract eyelid topological features, and to predict subtypes of levator function, using deep learning method to extract blinking features, in order to provide new ideas and means to assess eyelid topology and kinetics.

ELIGIBILITY:
Inclusion Criteria:

1. normal volunteers without eyelid diseases
2. patients with blepharoptosis
3. patients with blepharospasm
4. patients with dry eye disease
5. patients with Graves' disease

Exclusion Criteria:

variable ptosis (e.g., myasthenia gravis), entropion, ectropion, enophthalmos, exophthalmos, strabismus, and abnormalities of pupil

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 normal volunteers without eyelid diseases 100 patients with blepharoptosis 100 patients with blepharospasm 100 patients with dry eye disease 100 patients with Graves' disease
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
one-dimensional parameters of eyelid topology | through study completion, 5 years
  Palpebral fissure length [Margin reflex distance 1, Margin reflex distance 2], Lid length [Upper lid length, Lower lid length], Multiple mid-pupil lid distances
two-dimensional parameters of eyelid topology | through study completion, 5 years
  Palpebral fissure area [Medial area, Corneal area, Lateral area]
subtypes of levator function | through study completion, 5 years
  Levator function is classified into three categories: good, fair and poor

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Ye, Hangzhou, Zhejiang, China